CLINICAL TRIAL: NCT06219057
Title: Unfolding the Wisdom Within: A Clinical Trial Assessing the Impact of a Compassion Based Psychotherapeutic Intervention for Adolescents Placed in Child-welfare-based Residential Care
Brief Title: Unfolding the Wisdom Within: CFT for Adolescents in Residential Care
Acronym: CFT_RYC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Rita Ramos Miguel, Principal Investigator, Master in clinical psychology, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020.05840.BD
Record Dates: First submitted 2023-12-14; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Adolescent Behavior; Adolescent - Emotional Problem
Keywords: child-welfare-based residential care; compassion-focused therapy; adolescence; clinical randomized trial
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Intervention Model Description: To attain this project's aims a longitudinal research will take place. Adolescents living in residential youth care will be invited to participate. According to a criteria of convenience, 15 adolescents will receive the intervention (experimental group) and 15 other adolescents will receive the care as usual (control group).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Group of adolescents living in residential youth care. Participants selection will take as inclusion criteria: age (between 14 and 18 years old) and being placed in residential care at least for 1-month (allowing for an adjustment period); as exclusion criteria: a) cognitive impairment; b) psychotic symptoms; d) remaining in residential care less than 9-months, considering the study's length. They will be asked to fill in the self-report protocol at 3 different time points (baseline, post-test and 6-month follow-up).
  Intervention comprises the psychological intervention program "The Wise Adolescent", twenty individual psychotherapeutic sessions based on Compassion Focused Therapy.
  Interventions: Behavioral: The Wise Adolescent
- Care as Usual (No Intervention): Group of adolescents living in residential youth care. Participants selection will take as inclusion criteria: age (between 14 and 18 years old) and being placed in residential care at least for 1-month (allowing for an adjustment period); as exclusion criteria: a) cognitive impairment; b) psychotic symptoms; d) remaining in residential care less than 9-months, considering the study's length. They will be asked to fill in the self-report protocol at 3 different time points (baseline, post-test and 6-month follow-up).
  Participants in the control group will receive care as usual (TAU). There will be no restrictions on the care that can be provided and it may comprise no treatment or, instead, referral to a variety of health care professionals (e.g. psychologist, psychiatrist) with diverse dosage. TAU will be recorded in terms of timing and nature of any intervention received.

INTERVENTIONS:
Behavioral: The Wise Adolescent — The program encompasses 20 individual weekly sessions manualized. Its main objective is to help adolescents to create affiliative feelings towards themselves and to develop a more compassionate inner voice. Sessions are organized across 6 main domains: (1) placing ourselves in the challenges of life: evolutionary roots of our mind, how social circumstances and life experiences shape us; the 3-affect regulation systems; (2) understanding difficulties: compassion focused therapy case formulation; (3) understanding compassion: the three flows of compassion, its three pillars (caring commitment, wisdom, strength and courage); (4) compassionate mind training: cultivating the compassion skills (compassionate attention, imagery, reasoning, and behavior); (5) working with difficulties: fears, blocks and resistances to compassion; multiple selves; shame and self-criticism; (6) sustaining a compassionate mind: reviewing the gains and relapse prevention.
  Arms: Intervention

SUMMARY:
Residential care youth show extensive mental health intervention needs due to history of maltreatment and embedded characteristics of residential placement, leading to harmful and cumulative effects throughout development, linked to internalizing and externalizing difficulties. However, existing interventions show limited suitability and poor randomized effectiveness evaluation.

To overcome these shortcomings, a new compassion-based program for adolescents in residential care will be developed. A non-randomized trial will be run, testing the program´s effects over adolescents' psychological functioning and investigating whether changes in compassion are associated with changes over time in mental health difficulties. The moderator effect of age, gender and maltreatment history will be investigated.

Findings intend to: improve mental-health of youth in residential care, provide an evidence-based intervention to be delivered in residential care settings, increase empirical support of compassion-based interventions, amplifying its scope of delivery.

DETAILED DESCRIPTION:
Youth in residential care (YRC) are considered a vulnerable population, presenting higher levels of emotional and behavioural problems than normative peers. YRC exhibit a higher pooled prevalence for any mental disorder (49%) than the general children and adolescent population (13.4%). In Portugal, around 6118 youth are placed in residential care (55% of whom are adolescents), 89% due to history of maltreatment (HM) (neglect and psychological, physical and sexual abuse).

Residential care commonly occurs after a HM which, per se, plays an important role in predicting internalizing (e.g. anxiety, depression), externalizing (e.g. poor impulse control, aggression), and emotion regulation difficulties. HM also contributes to high levels of shame (the affective experience of feeling defective, undesirable) and self-criticism (negative self-evaluations which comprise condemning, attacking and judgemental thoughts directed to the self). Furthermore, although residential care is an attempt to provide protection and care, it frequently represents the loss of attachment figures, repeated moving placements, a less home-like environment and less individualized caregiving. Thus, it is essential that YRC receive interventions that counteract these vulnerabilities. Existing programs address mostly behavioural and cognitive domains, however: a) they are aimed primarily at fostering parental skills of caregivers, not fully meeting adolescents' developmental needs, b) they have limited randomized effectiveness evaluation, and c) findings do not show positive effects on attachment security or placement disruption.

Compassion-based interventions have been gaining growing empirical support in treating several mental health problems and have been shown to be suitable for children, adolescents, and adults. Previous research also demonstrated the benefits of targeting compassion related variables in the treatment of childhood maltreatment survivors, mitigating the association between childhood maltreatment and later emotion regulation difficulties.

Compassion is a motivation comprising a deep awareness regarding the suffering of one-self and others, tied to a wish and effort to relieve it. It is linked to healthy psychological functioning and quality of life. Additionally, compassion negatively predicts emotion regulation difficulties shame and self-criticism, as well as psychopathological problems.

The majority of available findings relates to adult samples, but empirical evidence suggests that compassionate mind training may also be well-timed for adolescents. Within adolescents' studies, compassion has been identified as revealing a buffering effect against psychological distress, partially mediating the relationship between victimization and psychological maladjustment. Differences on gender and age seem to be significant, with males and high school students reporting greater levels of compassion. Intervention studies have also provided support for compassion as a protective factor. Compassion training with adolescents in the community predicted reduction in negative affect, perceived stress, and depressive and anxiety symptoms.

In sum, YRC show wide mental health intervention needs that demand tailored interventions. Since the existing interventions showed limited randomized clinical effectiveness and considering the promising results of compassion based-interventions, the present research aims to broaden the spectrum of therapeutic care, developing and assessing the efficacy of a compassionate-based intervention specifically designed to address the needs from YRC.

ELIGIBILITY:
Inclusion Criteria:

1) Being placed in residential care at least for 1-month (allowing for an adjustment period)

Exclusion Criteria:

1. Cognitive impairment (assessed through a clinical interview; MINI-KID);
2. Presence of psychotic symptoms or suicidal ideation (according to the MINI-KID).

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-25 (Estimated); Study Completion 2024-08-03 (Estimated)

PRIMARY OUTCOMES:
Other as Shamer Scale - Short Adolescent version | Baseline, assessment 6-months after baseline; assessment 12-months after baseline
  The Other as Shamer Scale - Short Adolescent version comprises 8 items combined in one-factor measurement model that assesses a subject's perception of being negatively judged by others (i.e., external shame). Each item is rated on a five-point Likert scale reporting how frequently one experiences the feelings described in each statement (0 = never to 4 = almost always). Cronbach's alphas in the original version were .82 and good concurrent and divergent validity was showed. The Portuguese version reply the short version and presented an internal consistency of .90.
  Vagos, P., Ribeiro da Silva, D., Brazão, N., Rijo, D., & Gilbert, P. (2016). Dimensionality and measurement invariance of the Other as Shamer Scale across diverse adolescent samples. Personality and Individual Differences, 98, 289-296. http://dx.doi.org/10.1016/j.paid.2016.04.046
Forms of Self-Criticising and Self-Reassuring Scale | Baseline, assessment 6-months after baseline; assessment 12-months after baseline
  The Forms of Self-Criticising and Self-Reassuring Scale is a 22-item scale that measures two forms of self-criticism: (1) inadequate self, which focuses on a sense of personal inadequacy and (2) hated self, which assesses the desire to hurt or persecute the self. The scale also assesses self-reassurance. Items are rated on a five-point Likert scale (ranging from 0 = not at all like me to 4 = extremely like me).The original version of the scale presented good psychometric properties, with alphas of .90 for inadequate self and .86 for hated self and self-reassure. In the Portuguese version, internal consistency values were .89 for inadequate self, .80 for hated self, and .86 for self-reassure.
  Gilbert, P., Clark,M., Hempel, S.,Miles, J. N. V., & Irons, C. (2004). Criticising and reassuring oneself: An exploration of forms, styles and reasons in female students. British Journal of Clinical Psychology, 43(1), 31-50. https://doi.org/10.1348/014466504772812959
Compass of Shame Scale - adolescents version (COSS) | Baseline, assessment 6-months after baseline; assessment 12-months after baseline
  COSS assesses shame-coping styles. It includes 48 items, distributed over 12 scenarios assessing maladaptive coping styles: (1) Avoidance ( "I act as if it isn't so"); (2) Attack-Self ("I get mad at myself for not being good enough"); (3) Withdrawal ("I withdraw from the activity"); and (4) Attack-Other ("I get irritated with other people"). It also includes 10 items about adaptive responses to a shameful event (e.g., "When I feel lonely or left out, I talk to a friend"). All items in a five-point frequency scale (0 = never to 4 = almost always). The scale showed good and satisfactory internal consistency across all subscales (from α = .72 to α = .88
  Vagos, P., Ribeiro da Silva, D., Brazão, N., Rijo, D., & Elison, J. (2018). Psychometric properties of the compass of shame scale: Testing for measurement invariance across community boys and boys in foster care and juvenile detentions facilities. Child & Youth Care Forum, 48(1), 93-110. https://doi.org/10.1007/s10566-018-9474-x

SECONDARY OUTCOMES:
Self-compassion Scale | Baseline, assessment 6-months after baseline; assessment 12-months after baseline
  The Self-compassion Scale addresses self-compassion and instructs participants to answer its 26 self-reported items, rated in a five-point Likert-scale (ranging from 1 = almost never to 5 = almost always), regarding "how I typically act towards myself in difficult times". The scale has a total score and 6 subscales (Self-Kindness; Self-Judgement; Common Humanity; Isolation; Mindfulness; and Over-Identification). In the original version the total score showed very good internal consistency (α = .92) and the six subscales ranged from .75 to .81. In the Portuguese adolescent version, the total score had an internal consistency of .88 and the six subscales ranged from .70 to .79.
  Cunha, M., Xavier, A., & Castilho, P. (2015). Understanding self-compassion in adolescents: Validation study of the Self-Compassion Scale. Personality and Individual Differences, 93, 56-92. https://doi.org/10.1016/j.paid.2015.09.023
Compassion Scale | Baseline, assessment 6-months after baseline; assessment 12-months after baseline
  The Compassion Scale is a self-report instrument designed to measure compassion for others. This scale has 16 items rated on a 5-point Likert scale (from 1 to 5 points). The adolescent version showed adequacy of a hierarchical-CFA measurement model, with a general score of compassion and four specific factors (i.e., Kindness, Common Humanity, Mindfulness and Indifference). It also showed good internal reliability and construct validity.
  Pommier, E., Neff, K. D. & Tóth-Király I. (2019). The development and validation of the Compassion Scale. Assessment, 21-39.
Fears of Compassion Scales - Adolescents version | Baseline, assessment 6-months after baseline; assessment 12-months after baseline
  The Fears of Compassion Scales - Adolescents version (FCS-A) assesses fear of compassion for self, fear of compassion for others, and fear of compassion from others. It identifies barriers to giving compassion to oneself (15 items), to others (10 items), and receiving compassion from others (13 items). The items are rated on a five-point Likert scale (0 = don't agree at all to 4 = completely agree). The higher the score, the greater the one's fears, blocks and resistances to compassion. These scales showed good reliability with Cronbach's alpha's of .92 for self, .85 from others, and .84 for others in a student sample.
  Gilbert, P., McEwan, K., Matos, M., Rivis, A. (2011). Fears of compassion: Development of three self-report measures. Psychology and Psychotherapy: Theory, Research and Practice, 84, 239-255. https://doi.org/10.1348/147608310X526511
Social Safeness and Pleasure Scale - Adolescent version | Baseline, assessment 6-months after baseline; assessment 12-months after baseline
  Social Safeness and Pleasure Scale - Adolescent version is a unidimensional self-report questionnaire, composed of 11-items. It assesses how people interpret their social world as safe, soothing and warm (e.g., "I feel a sense of warmth in my relationships with people"). Participants rate each item using a five-point scale (1 = almost never to 5 = almost all the time); so, the total score of SSPS-A range from 11 to 55. In the original study, the SSPS achieved very good internal consistency (α = .91). The adolescent version achieved excelent internal consistency values (α > .93) and evidence for construct validity in relation to external variables was found.
  Miguel, R. R., Sousa, R., Santos, L., Brazão, N., Rijo, D., Castilho, Gilbert, P. (2022). Dimensionality and measurement invariance of the Social Safeness and Pleasure Scale in adolescents from community and residential youth care. Child Abuse and Neglect, 131, 105690. https://doi.org/10.1016/j.chiabu.2022.105690
Cognitive Emotion Regulation Questionnaire - Kids version (CERQ) | Baseline, assessment 6-months after baseline; assessment 12-months after baseline
  CERQ-Kids is a self-report questionnaire assessing cognitive emotional regulation strategies when facing stressful events. Its 36 items are spread across nine subscales: Self-Blame, Rumination, Positive Refocusing, Planning, Other-Blame, Catastrophizing, Putting into Perspective, Positive Reappraisal, and Acceptance. Each subscale has 4 items, answered on a five-point Likert scale that ranges from 1 (almost never) to 5 (almost always). The original version showed Cronbach's alpha ranging between 0.65 and 0.80. The Portuguese version proved to be a psychometrically adequate with alphas ranged between 0.62 and 0.87.
  Moreira, H., Vagos, P., Pereira, J., Fonseca, A., Canavarro, M. C., & Rijo, D. (2020). Psychometric properties of the Portuguese version of the cognitive emotion regulation questionnaire - kids version (CERQ-kids) among a sample of children and adolescents exposed to wildfires. Currently Psychology, 41, 2574-2585. https://doi.org/10.1007/s12144-020-00778-1
Kidscreen-10 index | Baseline, assessment 6-months after baseline; assessment 12-months after baseline
  Kidscreen-10 is a self-report measure assessing children's perception of their quality of life. It is a 10-item unidimensional questionnaire, answered using a five-point Likert scale that ranges from 1 (never; not at all) to 5 (always; extremely). The original version presented adequate reliability (α = .82) and temporal stability (ICC = .70) and demonstrated good criterion and construct validity. The Portuguese version confirmed the original unidimensional structure and showed adequate reliability (α = .78).
  Matos, M. G., Gaspar, T., & Simões, C. (2012). Health-related quality of life in Portuguese children and adolescents. Psicologia: Reflexão e Crítica, 25(2), 230-237. https://doi.org/10.1590/S0102- 79722012000200004
Depression, Anxiety and Stress Scale | Baseline, assessment 6-months after baseline; assessment 12-months after baseline
  Depression, Anxiety and Stress Scale is a self-report measure composed by 21 items assessing three dimensions of psychopathological symptoms: depression, anxiety, and stress. Items are rated using a four-point Likert scale for frequency (ranging from 0 = Does not apply to me at all to 3 = Applied to me very much or most of the time). Original version presented good internal consistency values for the three measures (α ≥ .84) as well the Portuguese version (α ≥ .74).
  Lovibond, P., & Lovibond, H. (1995). The structure of negative emotional states: Comparison of the depression anxiety stress scales (DASS) with Beck depressive and anxiety inventories. Behaviour Research and Therapy, 3, 335-343. https://doi.org/10.1016/0005-7967(94)00075-U
  Salvador, M.C., & Pires, C. (2020). Depression, Anxiety and Stress Scale: Psychometric properties in a Portuguese adolescent sample. Manuscript in preparation.
Achenbach System of Empirically Based Assessment | Baseline, assessment 6-months after baseline; assessment 12-months after baseline
  Achenbach System of Empirically Based Assessment describe a broad of emotional and behavioral problems in children and adolescents. Multicultural norms have been constructed. Informants rate the problem items as 0 = not true, 1 = somewhat or sometimes true, or 2 = very true or often true, over a period of 6 months.
  Two instruments were administered: (1) Youth self-report (YSR), a psychometric tool that assesses self-reported behavioral and emotional problems and the psychosocial competencies of adolescents between the ages of 11 and 18 years old.
  (2) Child Behavior Checklist (CBCL) was asked to be filled by the caregivers in the care institution.
  Achenbach, T. M. (2009). The Achenbach system of empirically based assessment (ASEBA): Development, findings, theory, and applications. Burlington: University of Vermont, Research Center for Children, Youth, and Families.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Miguel, Master, Principal Investigator — University of Coimbra, Portugal
Locations (1):
- Center for Research in Neuropsychology and Cognitive and Behavioral Intervention (CINEICC), Faculty of Psychology and Educational Sciences - University of Coimbra, Coimbra, Portugal

REFERENCES:
- [Background] [1] Campos, J., Barbosa-Ducharne, M., Dias, P., Rodrigues, S., Martins, A., & Leal, M. (2019). Emotional and behavioral problems and psychosocial skills in adolescents in residential care. Child and Adolescent Social Work Journal, 36, 237-246. https://doi.org/10.1007/s10560-018-0594-9
- [Background] [2] Haggman-Laitila, A., Salokekkila, P., & Karki, S. (2019). Young people's preparedness for adult life and coping after foster care: A systematic review of perceptions and experiences in the transition period. Child & Youth Care Forum, 48, 633-661. https://doi.org/10.1007/s10566-019-09499-4
- [Background] Bronsard G, Alessandrini M, Fond G, Loundou A, Auquier P, Tordjman S, Boyer L. The Prevalence of Mental Disorders Among Children and Adolescents in the Child Welfare System: A Systematic Review and Meta-Analysis. Medicine (Baltimore). 2016 Feb;95(7):e2622. doi: 10.1097/MD.0000000000002622. PMID 26886603
- [Background] Polanczyk GV, Salum GA, Sugaya LS, Caye A, Rohde LA. Annual research review: A meta-analysis of the worldwide prevalence of mental disorders in children and adolescents. J Child Psychol Psychiatry. 2015 Mar;56(3):345-65. doi: 10.1111/jcpp.12381. Epub 2015 Feb 3. PMID 25649325
- [Background] [5] Departamento de Desenvolvimento Social. (2019). Casa 2018 - Relatório de caracterização anual da situação de acolhimento das crianças e jovens [Annual report on the characterization of youth in out-of-home placement]. Portugal, Instituto da Segurança Social, I.P. http://www.seg-social.pt/documents/10152/16662972/Relat%C3%B3rio_CASA2018/f2bd8e0a-7e57-4664-ad1e-f1cebcc6498e
- [Background] Li M, D'Arcy C, Meng X. Maltreatment in childhood substantially increases the risk of adult depression and anxiety in prospective cohort studies: systematic review, meta-analysis, and proportional attributable fractions. Psychol Med. 2016 Mar;46(4):717-30. doi: 10.1017/S0033291715002743. Epub 2015 Dec 28. PMID 26708271
- [Background] Norman RE, Byambaa M, De R, Butchart A, Scott J, Vos T. The long-term health consequences of child physical abuse, emotional abuse, and neglect: a systematic review and meta-analysis. PLoS Med. 2012;9(11):e1001349. doi: 10.1371/journal.pmed.1001349. Epub 2012 Nov 27. PMID 23209385
- [Background] Heleniak C, Jenness JL, Stoep AV, McCauley E, McLaughlin KA. Childhood Maltreatment Exposure and Disruptions in Emotion Regulation: A Transdiagnostic Pathway to Adolescent Internalizing and Externalizing Psychopathology. Cognit Ther Res. 2016 Jun;40(3):394-415. doi: 10.1007/s10608-015-9735-z. Epub 2015 Dec 12. PMID 27695145
- [Background] Michl LC, Handley ED, Rogosch F, Cicchetti D, Toth SL. Self-Criticism as a Mechanism Linking Childhood Maltreatment and Maternal Efficacy Beliefs in Low-Income Mothers With and Without Depression. Child Maltreat. 2015 Nov;20(4):291-300. doi: 10.1177/1077559515602095. Epub 2015 Aug 27. PMID 26318693
- [Background] Shahar B, Doron G, Szepsenwol O. Childhood Maltreatment, Shame-Proneness and Self-Criticism in Social Anxiety Disorder: A Sequential Mediational Model. Clin Psychol Psychother. 2015 Nov-Dec;22(6):570-9. doi: 10.1002/cpp.1918. Epub 2014 Sep 5. PMID 25196782
- [Background] Li D, Chng GS, Chu CM. Comparing Long-Term Placement Outcomes of Residential and Family Foster Care: A Meta-Analysis. Trauma Violence Abuse. 2019 Dec;20(5):653-664. doi: 10.1177/1524838017726427. Epub 2017 Aug 31. PMID 29333987
- [Background] [12] Nobre Lima, L. (2009). Estórias e projetos de vida de adolescentes institucionalizados [Stories and life projects from residential care adolescents] (Unpublished doctoral dissertation). (Unpublished doctoral dissertation). Faculty of Psychology and Educational Sciences, University of Coimbra, Coimbra, Portugal.
- [Background] Hambrick EP, Oppenheim-Weller S, N'zi AM, Taussig HN. Mental Health Interventions for Children in Foster Care: A Systematic Review. Child Youth Serv Rev. 2016 Nov;70:65-77. doi: 10.1016/j.childyouth.2016.09.002. Epub 2016 Sep 8. PMID 28496286
- [Background] Schoemaker NK, Wentholt WGM, Goemans A, Vermeer HJ, Juffer F, Alink LRA. A meta-analytic review of parenting interventions in foster care and adoption. Dev Psychopathol. 2020 Aug;32(3):1149-1172. doi: 10.1017/S0954579419000798. PMID 31366418
- [Background] Kirby JN, Tellegen CL, Steindl SR. A Meta-Analysis of Compassion-Based Interventions: Current State of Knowledge and Future Directions. Behav Ther. 2017 Nov;48(6):778-792. doi: 10.1016/j.beth.2017.06.003. Epub 2017 Jun 21. PMID 29029675
- [Background] [16] Gilbert, P., & Procter, S. (2006). Compassionate mind training for people with high shame and self-criticism: Overview and pilot study of a group therapy approach. Clinical Psychology and Psychotherapy, 13, 353-379. http://dx.doi.org/10.1002/cpp.507
- [Background] [17] Vettese, L.C., Dyer, C.E., Li, W.L., & Wekerle, C. (2011). Does self-compassion mitigate the association between childhood maltreatment and later emotion regulation difficulties? A preliminary investigation. International Journal of Mental Health and Addiction, 9, 480-491. http://dx.doi.org/10.1007/s11469-011-9340-7
- [Background] Zessin U, Dickhauser O, Garbade S. The Relationship Between Self-Compassion and Well-Being: A Meta-Analysis. Appl Psychol Health Well Being. 2015 Nov;7(3):340-64. doi: 10.1111/aphw.12051. Epub 2015 Aug 26. PMID 26311196
- [Background] Finlay-Jones AL, Rees CS, Kane RT. Self-Compassion, Emotion Regulation and Stress among Australian Psychologists: Testing an Emotion Regulation Model of Self-Compassion Using Structural Equation Modeling. PLoS One. 2015 Jul 24;10(7):e0133481. doi: 10.1371/journal.pone.0133481. eCollection 2015. PMID 26207900
- [Background] MacBeth A, Gumley A. Exploring compassion: a meta-analysis of the association between self-compassion and psychopathology. Clin Psychol Rev. 2012 Aug;32(6):545-52. doi: 10.1016/j.cpr.2012.06.003. Epub 2012 Jun 23. PMID 22796446
- [Background] Bluth K, Gaylord SA, Campo RA, Mullarkey MC, Hobbs L. Making Friends With Yourself: A Mixed Methods Pilot Study of a Mindful Self-Compassion Program for Adolescents. Mindfulness (N Y). 2016 Mar 1;7(2):479-492. doi: 10.1007/s12671-015-0476-6. Epub 2015 Dec 19. PMID 27110301
- [Background] [22] Carona, C., Rijo, D., Salvador, C., Castilho, P. & Gilbert, P. (2017). Compassion-focused therapy with children and adolescents. BJPsych Advances, 23(4), 240-252. http://dx.doi.org/10.1192/apt.bp.115.015420
- [Background] [23] Ribeiro da Silva, D., Rijo, D., Salekin, R. T., Paulo, M., Miguel, R., & Gilbert, P. (2020). Clinical change in psychopathic traits after the PSYCHOPATHY.COMP program: Preliminary findings of a controlled trial with male detained youth. Journal of Experimental Criminology. https://doi.org/10.1007/s11292-020-09418-x
- [Background] [24] Salvador, C., Carona, C., Catilho, P. & Rijo, D. (2017). Self-criticism and self-compassion in adolescents: Two forms of self-relating and their implications for psychopathology and treatment. Turkiye Klinikleri Child Psychiatry -Special Topics, 3(2):132-8.
- [Background] Jativa R, Cerezo MA. The mediating role of self-compassion in the relationship between victimization and psychological maladjustment in a sample of adolescents. Child Abuse Negl. 2014 Jul;38(7):1180-90. doi: 10.1016/j.chiabu.2014.04.005. Epub 2014 May 5. PMID 24811571
- [Background] [26] Yarnell, L. M., Stafford, R. E., Neff, K. D., Reilly, E. D., Knox, M. C., & Mullarkey, M. (2015). Meta-analysis of gender differences in self-compassion. Self and Identity, 14(5), 499-520. https://doi.org/10.1080/15298868.2015.1029966
- [Background] Bluth K, Eisenlohr-Moul TA. Response to a mindful self-compassion intervention in teens: A within-person association of mindfulness, self-compassion, and emotional well-being outcomes. J Adolesc. 2017 Jun;57:108-118. doi: 10.1016/j.adolescence.2017.04.001. Epub 2017 Apr 14. PMID 28414965